CLINICAL TRIAL: NCT01432626
Title: The Evaluation of the Pathogenesis of Stress-Induced Cardiomyopathy by I-123 MIBG Imaging
Brief Title: Pathogenesis of Stress-Induced Cardiomyopathy by I-123 MIBG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: GE Healthcare (Industry)
Responsible Party: Principal Investigator, Prem Soman, Principle Investigator, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PRO10080198
Record Dates: First submitted 2011-09-07; First posted 2011-09-13 (Estimated); Results first posted 2016-03-22 (Estimated); Last update posted 2016-03-22 (Estimated); Status verified 2016-03

CONDITIONS: Stress Induced Cardiomyopathy
Keywords: stress induced cardiomyopathy; broken heart syndrome; Takotsubo cardiomyopathy; transient apical ballooning syndrome; apical ballooning cardiomyopathy; stress cardiomyopathy; non-ischemic cardiomyopathy
MeSH Terms: conditions — Takotsubo Cardiomyopathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Stress Induced Cardiomyopathy Patients (Experimental): Patients presenting with stress induced cardiomyopathy, after meeting the Mayo criteria (normal coronary anatomy, EKG changes/Enzyme abnormalities, wall motion abnormalities consistent with stress induced cardiomyopathy and no evidence of pheochromocytoma) and signing informed consent, will receive an I123-mIBG scan to determine the sympathetic function of the heart during the acute presentation and after functional recovery.
  Interventions: Drug: I-123 radiolabeled metaiodobenzylguanidine cardiac imaging

INTERVENTIONS:
Drug: I-123 radiolabeled metaiodobenzylguanidine cardiac imaging — All subjects will receive an intravenous injection of 10 mCi (370 MBq) of 123I-mIBG. A ±10% tolerance of the nominal dose will be allowed, thus yielding an acceptable dose range of 9 to 11 mCi (333 to 407 MBq). The investigational medicinal product will be administered in a volume of 5 mL (diluted using 0.9% sodium chloride as needed) and injected over 1 to 2 minutes. The patient will have planar and SPECT imaging performed after the dose is administered. This dosing and imaging procedure will be performed during the acute phase and after the patient has recovered cardiac function, approximately 6 weeks later. This means that each study subject will receive a total of 2 doses of I123-mIBG at 2 different time points.
  Other Names: AdreVeiw

SUMMARY:
Objective: The objective of this pilot study is to characterize the cardiac uptake patterns of I-123 mIBG in stress-induced (Takotsubo's) cardiomyopathy.

Hypothesis: Perturbations in sympathetic innervation are the underlying pathogenesis of stress induced cardiomyopathy and will result in abnormalities in I-123 mIBG cardiac imaging. Thus, planar and SPECT I-123 MIBG imaging will provide insight into the pathogenesis of stress-induced cardiomyopathy, and may lead to the development of more specific diagnostic criteria.

Study design: This proposal is for a prospective pilot study to characterize perturbations in cardiac sympathetic innervation in patients with stress induced cardiomyopathy by performing planar and SPECT I-123 MIBG imaging during the acute presentation and after recovery of LV function.

DETAILED DESCRIPTION:
Background: Since the initial Japanese description of Takotsubo's cardiomyopathy in 1991 as a transient systolic dysfunction of the apical or mid left ventricular segments in the absence of obstructive coronary artery disease, stress induced cardiomyopathy has been increasingly recognized in the Unites States. Takotsubo's cardiomyopathy accounts for 1.2 to 2.2 percent of all cases of acute coronary syndrome. The current American Heart Association Statistical Update estimates that approximately 1.2 million Americans will experience an acute coronary event in 2010. Based on this estimate, between 15 and 26 thousand Americans will have stress induced cardiomyopathy annually. Takotsubo's cardiomyopathy has also been described in stroke and critically ill patients. Post menopausal women are disproportionally affected, accounting for 80 to 100 percent of the patient population. These patients classically present with signs of acute heart failure or acute coronary syndrome after a severe emotional stress. The presentation may include chest pain, shortness of breath, elevated troponin enzymes, ST segment elevations, deep T-wave inversions, ventricular arrhythmias, pulmonary edema or elevated biomarkers. Cardiac catheterization reveals angiographically normal coronary arteries while the ventriculogram and the echocardiogram shows apical ballooning with basal hyperkinesis. While the majority of patients recover complete function within few days to two weeks, up to eight percent of the patients will die from the acute heart failure.

The etiology of stress-induced cardiomyopathy remains speculative. Catecholamine excess leading to microvascular dysfunction or direct cardiomyocyte toxicity is hypothesized as the most likely etiology. This hypothesis is supported by the fact that most patients with Takotsubo's cardiomyopathy experience an intense physical or emotional stress. Furthermore, several other observations support this hypothesis. First, catecholamines levels are elevated in patients with stress induced cardiomyopathy at presentation when compared to patients with acute coronary syndrome. Second, multi-vessel coronary vasospasm and transient myocardial perfusion defects have been identified repeatedly in this population. Third, myocardial biopsies show myocarditis, interstitial fibrosis and mononuclear infiltrates, signs consistent with catecholamine toxicity. Fourth, in a mouse model, elevated epinephrine levels cause a switch from beta-2 adrenoreceptor mediated Gs protein signaling to Gi protein signaling, which is negatively inotropic. These findings all support the theory that there is altered sympathetic activity in patients with stress induced cardiomyopathy.

Thus, based on the existing knowledge base of this intriguing disease, an imaging approach that specifically evaluates the sympathetic activation state of the myocardium would appear to be ideally suited to further explore pathophysiology. I-123 radiolabeled metaiodobenzylguanidine, (mIBG) imaging allows for direct analysis of cardiac sympathetic function because it is structurally similar to norepinephrine (NE), and is transported into the cardiac sympathetic neurons by human norepinephrine transporter 1 ( hNET1), in the synaptic cleft. Unlike NE, mIBG is not metabolized by monoamine oxidase or catechol-o-methyl transferase. mIBG requires an intact myocardial sympathetic nervous system for uptake, is stored in the presynaptic vesicles and is released by stimulation with acetylcholine. Experimental manipulation of cardiac sympathetic function alters mIBG uptake and distribution. Planar imaging acquisition enables evaluation of sympathetic activation, while SPECT characterizes regional abnormalities. Measurement of the heart to mediastinal ratio during early and delayed planimetry assesses the initial uptake and washout of the tracer. mIBG uptake follows one of three general patterns: good uptake and retention, good uptake with washout or poor uptake. The different patterns likely represent the level of sympathetic activation, increase in sympathetic tone and heart failure-induced damage to the myocardial sympathetic nervous system. mIBG uptake is altered in patient with diabetic neuropathy, congestive heart failure, myocardial infarction. The uptake and washout patterns correlate with severity of neuropathy, severity of congestive heart failure, congestive heart failure treatment response, improvement in ejection fraction, cardiac death and ventricular arrhythmogenic potential.

Preliminary data in patients with Takotsubo's cardiomyopathy has shown decrease in mIBG uptake with an increased washout in the acute phase, with improved retention after left ventricular functional recovery. Furthermore, regional decrease in tracer uptake corresponds to the regional wall motion abnormalities. However, a systematic exploration of mIBG uptake patterns in consecutive patients with Takotsubo's cardiomyopathy has not been performed. Of note, PET imaging with 11C Hydroxyephedrine has described similar sympathetic dysfunction in Takotsubo's cardiomyopathy.

ELIGIBILITY:
Inclusion Criteria:

* The subject is ≥18 years of age at study entry.
* The subject is able and willing to comply with study procedures and signed and dated informed consent is obtained.
* The subject is male, or a female who is either surgically sterile (has a documented bilateral oophorectomy and/or hysterectomy), postmenopausal (cessation of menses for more than 1 year), non-lactating, or of childbearing potential for whom the result of a urine pregnancy test performed at screening is negative.
* The subject's left heart catheterization (obtained as part of the clinical evaluation) is without clinically significant coronary atherosclerotic disease.
* The subject's echocardiogram (obtained as part of the clinical evaluation) is consistent with a diagnosis of Takotsubo's Cardiomyopathy.
* The patient's electrocardiogram or cardiac enzymes including troponin or CKMB (obtained as part of the clinical evaluation) is abnormal.
* The patient does not have a diagnosis or suspicion of Pheochromocytoma.

Exclusion Criteria:

* The subject has previously received I123-MIBG or I131-MIBG.
* The subject has a ventricular pacemaker that routinely functions (>5% paced beats) or has received defibrillation (either external or via an ICD), anti-tachycardic pacing, or cardioversion to treat a previous arrhythmic event.
* The subject was previously entered into this study or has participated in any other investigational medicinal product or medical device study within 30 days of enrollment.
* The subject has a previous history or suspicion of significant allergic reaction or anaphylaxis to iodine or iodinated compounds.
* The subject had cardiac revascularization (eg, percutaneous transluminal coronary angioplasty, PCI, or CABG) or insertion of an ICD within the last 30 days.
* The subject has a serious non-cardiac medical condition associated with significant elevation of plasma catecholamines including Pheochromocytoma.
* The subject is claustrophobic or has a movement disorder that prevents him/her from lying still in a supine position for up to an hour at a time.
* The subject has renal insufficiency (serum creatinine > 3.0 mg/dl [265umol/L]).
* The subject has participated in a research study using ionizing radiation in the previous 12 months.
* The subject has a history of Type I or Type II Diabetes Mellitus with signs of neurological involvement, signs or symptoms of neurological disease (eg, Parkinson's Disease, Multiple System Atrophy, Parkinsonian syndromes), or other diseases known to affect the sympathetic nervous system.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2011-09; Primary Completion 2014-12 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Prem Soman, MD, Principal Investigator — University of Pittsburgh Heart Vascular Institute
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Stress Induced Cardiomyopathy Patients: Patients with stress induced cardiomyopathy, by the Mayo criteria (normal coronary anatomy, EKG changes/Enzyme abnormalities, wall motion abnormalities consistent with stress induced cardiomyopathy and no evidence of pheochromocytoma) and signing informed consent, will receive an I123-mIBG scan to determine the sympathetic function of the heart during the acute presentation and after functional recovery.
  I-123 radiolabeled metaiodobenzylguanidine cardiac imaging: All subjects will receive an intravenous injection of 10 mCi (370 MBq) of 123I-mIBG. A ±10% tolerance of the nominal dose will be allowed, thus yielding an acceptable dose range of 9 to 11 mCi (333 to 407 MBq). The patient will have planar and SPECT imaging performed after the dose is administered. This dosing and imaging procedure will be performed during the acute phase and after the patient has recovered cardiac function, approximately 6 weeks later.
Period: Overall Study
Arm/Group | Stress Induced Cardiomyopathy Patients
Started | 10
Completed | 3 (Completed both images)
Not Completed | 7
Not completed — LV function recovered | 2
Not completed — Withdrawal by Subject | 2
Not completed — Only 1 image competed | 2
Not completed — Imaging agent not available | 1

BASELINE CHARACTERISTICS:
Arm/Group | Stress Induced Cardiomyopathy Patients
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Had an Abnormal Regional Uptake of I-123 mIBG at Baseline (Acute Phase) and the Number of Participants Who Had an Abnormal I-123 mIBG Uptake on Follow up (Recovery Phase)
Description: Number of participants who had an abnormal regional uptake of I-123 mIBG at baseline (acute phase) and the number of participants who had an abnormal I-123 mIBG uptake on follow up (recovery phase)
Time Frame: During the acute phase (2-5 days with an expected mean 3 days) and after recovery of cardiac function (6 weeks)
Measure: Number; unit: participants
Arm/Group | Stress Induced Cardiomyopathy Patients
Number analyzed (Participants) | 3
participants
  Abnormal at baseline (acute phase) | 3
  Abnormal at follow up (recovery phase) | 1

ADVERSE EVENTS:
Description: Only patients who had at least one scan (n=5) were exposed to any potential adverse events.
Arm/Group | Stress Induced Cardiomyopathy Patients
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No